CLINICAL TRIAL: NCT01674998
Title: Understanding Autonomic Function in REM Sleep Behavior Disorder, Parkinsonism and Controls
Brief Title: Understanding the Natural History of REM Sleep Behavior Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Parkinson's Institute (Other)
Responsible Party: Principal Investigator, J. William Langston, Founder and CEO, The Parkinson's Institute
Other Study IDs: 11-DAT-013
Record Dates: First submitted 2012-08-27; First posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: REM Sleep Behavior Disorder
Keywords: REM Sleep Behavior Disorder; RBD; Dream; Dreams
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and/or saliva DNA

SUMMARY:
The purpose of this research study is to determine if safe, simple and non-invasive tests such as an electrocardiogram (EKG), a smell test, or a blood test could be used to identify neurological disorders before typical symptoms occur. Researchers believe that early identification of these disorders could lead to treatments to prevent, delay, or slow the development of one of more of these diseases. Some people with REM sleep behavior disorder (RBD) may go on to develop Parkinson's disease or another related neurological disorder, but many do not.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic REM sleep behavior

Exclusion Criteria:

* Parkinson's disease
* Alzheimer's disease
* Multiple system atrophy
* Dementia
* Minors

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sleep disorders clinics Neurology practices Medical practices Sleep disorders support groups Web-based advertisements Community outreach
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-07

CONTACTS AND LOCATIONS:
Locations (1):
- The Parkinson's Institute, Sunnyvale, California, United States